CLINICAL TRIAL: NCT04741243
Title: Effect of Extracorporeal Shock Therapy for Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Shaimaa Mohamed Hamed (Unknown)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo Un 99
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was done by sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy (Experimental): was used for 15 minutes in a prone position for both groups (A&B) before the treatment. shock wave were used to heat small areas, and allow for decrease pain, muscle spasm, and provide vasodilatation of the blood vessels supplying the area
  Interventions: Device: Extracorporeal Shock wave
- dietary modification (Experimental): Dietary modifications are changes made during food preparation, processing, and consumption to increase the bioavailability of micronutrients-and reduce micronutrient deficiencies-in food at the commercial or individual/household level.
  Interventions: Device: Extracorporeal Shock wave

INTERVENTIONS:
Device: Extracorporeal Shock wave — Dietary modifications are changes made during food preparation, processing, and consumption to increase the bioavailability of micronutrients-and reduce micronutrient deficiencies-in food at the commercial or individual/household level
  Other Names: dietary modification

SUMMARY:
This study was carried out upon forty women diagnosed as primary dysmenorrhea. They were selected from outpatient clinics of gynecology of Ain Shams University Hospital, Cairo University. Their age ranged from 25-35 years, BMI<30kg/ m².

DETAILED DESCRIPTION:
Patients with primary dysmenorrhea diagnosed by a physician, spondylolisthesis and chronic low back pain were excluded from the study. They were randomly assigned into two equal groups (A& B). Group (A) consisted of twenty subjects, with an average age 29.2±1.9Yrs, and BMI 27.28±2.1kg/m2 who received Extracorporeal shock waves. Group (B) consisted of twenty patients, with an average age 28.58±2.2Yrs, and BMI 28.92±0.7kg/m2 who received sham technique. A hot pack was used for 15 minutes for both groups (A&B) before the treatment.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* forty virgin females.
* their age ranged between 25 to 35 years old.
* Body mass index (BMI) <30kg/ m².

Exclusion Criteria:

* females with pelvic pathology as endometriosis.
* females have irregular menstrual cycles.
* females have secondary dysmenorrhea.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | three months
  Visual analogue scale: that was used to determine the pain intensity level. It consists of 10 cm as a horizontal line with one end represented that (0= no pain) and the other end (10= worst pain). The assessment was performed for every woman in both groups (A, B) before and after the treatment program.

SECONDARY OUTCOMES:
analysis of circulating β-endorphin | three months
  assessment of circulating β-endorphin was done before and after the treatment progam

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — Cairo University
Locations (1):
- Ghada Elrefaye, Giza, Cairo Governorate, Egypt